CLINICAL TRIAL: NCT04549285
Title: A Phase I Pilot Study of the Safety of Infusions of Allogeneic Human Cord Tissue Mesenchymal Stromal Cells in Children With Multisystem Inflammatory Syndrome in Children (MIS-C)
Brief Title: Infusions of Mesenchymal Stromal Cells in Children With Multisystem Inflammatory Syndrome
Acronym: MISTIC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No accrual
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Jerome Harris Distinguished Professor of Pediatrics, Professor of Pathology; Director, Marcus Center for Cellular Cures; Director, Pediatric Blood and Marrow Transplant Program;, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106044
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Multisystem Inflammatory Syndrome in Children
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hCT-MSC infusion (Experimental): Doses will be given on days 1, 2, 3, and a fourth, optional dose may be given on day 7 at the discretion of the investigator and the treating physician.
  Interventions: Biological: Human Cord Tissue Mesenchymal Stromal Cells (hCT-MSCs)

INTERVENTIONS:
Biological: Human Cord Tissue Mesenchymal Stromal Cells (hCT-MSCs) — Human Umbilical Cord Tissue-derived Mesenchymal Stromal Cells (hCT-MSC):
  hCT-MSCs is an allogeneic cell product manufactured from donated umbilical cord tissue that is digested and expanded in culture, cryopreserved and banked. Doses contain 2x10^6 cells/kg (up to a maximum dose of 100x10^6 cells) diluted in plasmalyte-A with 5% HSA to a volume of 20-40mL.

SUMMARY:
The purpose of this multi-site, pilot study is to test whether infusions of human cord tissue mesenchymal stromal cells (hCT-MSC) are safe in children with multi system inflammatory syndrome (MIS-C). We will also describe the symptom course and duration of this hyper-inflammatory syndrome in these patients. Six patients less than 21 years old with MIS-C that is refractory to intravenous immune globulin (IVIG) and/or steroids will be given intravenous infusions of hCT-MSCs. Doses of 2x10^6 cells/kg (up to a maximum dose of 100x10^6 cells) will be given on days 1, 2, 3, +/-7 (day 7 is optional). Participants will be followed up to 90 days after administration for severe adverse events and survival. Safety will be evaluated through adverse event monitoring, clinical evaluations (i.e., vital signs, physical examinations), laboratory tests (i.e., hematology, serum chemistries, and urinalysis), and cardiac function (i.e., echocardiogram, ECG) from the signing of informed consent and throughout the patient's participation in this treatment protocol.

DETAILED DESCRIPTION:
This phase I, multisite, pilot study will test whether infusions of human cord tissue derived MSCs (hCT-MSC) are safe in children with multisystem inflammatory syndrome (MIS-C).

The study population will consist of six patients 18 to <21 years old with a life expectancy ≥ 72 hours and COVID-19 related MIS-C that is refractory to treatment with intravenous immune globulin (IVIG).

Multisystem inflammatory syndrome in children (MIS-C) is a newly recognized, serious, hyper-inflammatory syndrome that is occurring in small numbers of children, many of whom are within a month or so of recovering from a COVID-19 infection. While the clinical presentation varies, affected patients are typically previously healthy individuals who are less than 21 years of age. The diagnostic criteria include fever, laboratory evidence of inflammation, and multisystem involvement requiring hospitalization. Up to 75% of patients present with an element of cardiogenic shock requiring inotropic support, with some also requiring intubation with mechanical ventilation. Reported supportive treatments have included intravenous immune globulin (IVIG), tocilizumab, methylprednisolone, and aspirin. In the limited cases reported, up to 50% of children with MIS-C have antibodies to COVID-19 in their blood and may or may not be PCR positive on a nasal swab or throat culture. The disease is incompletely understood but currently believed, at least in part, to be a hyper-immune response to a recent COVID-19 infection.

In laboratory experiments, MSCs have been shown to inhibit T-cell proliferation and decrease production of pro-inflammatory cytokines. In animal models, up to 70% of infused cells are engulfed by lung macrophages, leading to secretion of anti-inflammatory molecules by these macrophages. These observations have led to the hypothesis that MSCs may work through both anti-inflammatory, immune-modulatory, and regenerative mechanisms.

Over the past several months, MSCs have been tested in small cohorts of adult patients with COVID-19 Acute Respiratory Distress Syndrome to determine if the cytokine storm hypothesized to cause this complication could be suppressed by MSCs. Early results are encouraging, and formal clinical trials are underway. Extending this work into the pediatric population, the hypothesis of this study is that infusion of hCT-MSC can reverse the pro-inflammatory state in children with MIS-C.

This is a 6 patient, multisite, pilot study to test whether infusions of hCT-MSC are safe in pediatric patients with MIS-C. Information will also be gathered about the duration and severity of the participant's multisystem inflammatory syndrome. hCT-MSCs will be manufactured at Duke University Medical Center in the Robertson GMP Cell Manufacturing Laboratory and shipped frozen to the treatment site, where they will remain stored in the vapor phase of liquid nitrogen until the day of dosing.

The baseline evaluation will include vital signs (heart rate, blood pressure, temperature, respiratory rate), echocardiogram, ECG or telemetry strip, HLA typing, Panel Reactive Antibody (anti-HLA antibody), inflammatory markers, blood counts, blood chemistry, coagulation, and COVID-19 PCR and antibody tests.Patients will be dosed with 2x10^6 hCT-MSCs/kg. Doses will be given on days 1, 2, 3, and a fourth, optional dose may be given on day 7 at the discretion of the investigator and the treating physician. Prior to the infusion, premedications (Benadryl, Hydrocortisone, 0.5mg/kg each) will be administered. The hCT-MSCs will be administered intravenously over 30-60 minutes via a syringe pump. Pulse oximetry will be monitored continuously throughout the infusion and IV fluids will be managed by the care team. Afterwards, the participant will continue to be monitored in their care setting per institutional standards. Participants will be evaluated by study staff the day after the infusion to assess for any infusion-related adverse reactions or complications.

The participant will be monitored by study staff to assess for any infusion related adverse reactions or complications until discharge. Additional follow-up will occur on days 14, 28, and 90. Follow up testing will include assessment for adverse events as well as the tests done at baseline (with the exception of HLA typing and COVID PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to <21 years
2. Diagnosis: must meet ALL below criteria for COVID-19 related MIS-C as defined by the CDC.

   1. Age <21 years
   2. No alternative plausible diagnoses
   3. Positive for current or recent SARS-CoV-2 infection or COVID-19 exposure within the 4 weeks prior to the onset of symptoms. Exposure may be measure by RT-PCR, Serology, Antigen test, or History.
   4. ALL of the following clinical symptoms:

      * Fever ≥38.0 degrees C for ≥24 hours or report of subjective fever lasting

        * 24 hours
      * Laboratory evidence of inflammation, including, but not limited to, one or more of the following: an elevated CRP, ESR, fibrinogen, procalcitonin, d- dimer, ferritin, LDH, or IL-6; elevated neutrophils, reduced lymphocytes, low albumin
      * Clinically severe disease that requires hospitalization
      * Multisystem (≥2) organ involvement:

      I. Cardiovascular involvement (ANY of the listed criteria):
      * Cardiac dysrhythmia or arrythmia (NOTE: patients with prolonged QT interval or unstable dys/arrythmias are not eligible)
      * Ejection fraction 35%-<55%
      * Pulmonary edema due to left heart failure
      * Pericarditis or pericardial effusion (not requiring drainage)
      * B-type natriuretic peptide (BNP) >400 pg/mL
      * Elevated troponin (based on the upper limit of normal for the laboratory running the assay)
      * Receipt of vasopressor or vasoactive support

      II. Respiratory Involvement (includes ANY of the listed criteria)
      * Receipt of mechanical ventilation or any type of supplemental oxygen (or increased support for patients receiving respiratory support at baseline)
      * Pulmonary infiltrates on chest radiograph
      * Lower respiratory infection
      * Pleural effusion (not requiring chest tube)
      * Pneumothorax (not requiring chest tube)

      III. Ophthalmologic involvement
      * Iritis or uveitis

      IV. Gastrointestinal involvement (includes ANY of the listed criteria)
      * Nausea/vomiting
      * Diarrhea
      * Abdominal pain
      * Pancreatitis (amylase and/or lipase >200 U/L or radiologic findings)
      * Hepatitis (AST and/or ALT >500 U/L)
      * Gallbladder hydrops or edema

      V. Hematologic involvement (includes ANY of the listed criteria)
      * Total white blood cell <4 x10^3/μL
      * Anemia (hemoglobin <9 g/dL)
      * Platelet count <150,000 /μL
      * Hemolysis VI. Mucocutaneous involvement (includes ANY of the listed criteria)
      * Bilateral conjunctival injection
      * Oral mucosal changes
      * Peripheral extremity changes
      * Rash or skin ulcers
      * 'COVID' toes
      * Swollen red cracked lips
      * Erythema of palms or soles
      * Edema of hands or feet
      * Periungual (nails) desquamation
      * Conjunctivitis
      * Peripheral gangrene

      VII. Musculoskeletal involvement (includes ANY of the listed criteria)
      * Arthritis or arthralgia involvement
      * Myositis or myalgia
3. Prior therapy: must have been treated with IVIG (maximum cumulative dose of 5g/kg) 1-7 days prior to enrollment. Patients will be eligible if they have progressive symptoms ≥24 hours after initiation of IVIG or lack of response ≥48 hours after initiation of IVIG. Lack of response is defined as inability wean off of supportive care measures (ie. vasopressors, mechanical ventilation, oxygen support) or lack of improvement in inflammatory markers.
4. Prior treatment with immunomodulators (e.g. tocilizumab, etc) is allowed if there was no response or progressive disease 2 days (48 hours) or more after initiation of this therapy.
5. Life expectancy ≥ 72 hours
6. Legal authorized representative consent

Exclusion Criteria:

1. Evidence of acquired or congenital immunodeficiency (due to immunosuppressive therapy, HIV, previous treatment for cancer, etc.)
2. History of cancer
3. History of previous treatments with MSCs or other cell therapies
4. Patient is enrolled in any other IND-sponsored clinical trials for COVID-19
5. Evidence of pregnancy or lactation
6. Moribund patient not expected to survive > 24 hours
7. Patient is receiving Extracorporeal Membrane Oxygenation (ECMO)
8. Patient received CPR for this condition
9. Patients who have acquired thrombotic risk due to COVID, e.g., VTE, pulmonary embolism, stroke, intracranial hemorrhage, ischemia of an extremity, or prone to thrombotic conditions, e.g., Factor V Leiden mutations, lupus anti-coagulant, etc.
10. Patients with history of DMSO allergies
11. ECG exclusions: prolonged QT interval, changes suggestive of myocardial ischemia, unstable cardiac dys/arrythmia that requires medical stabilization (ie.

    unstable supraventricular tachycardia, ventricular tachycardia, or ventricular fibrillation)
12. Echocardiogram exclusions: Dilated coronary artery(ies) (z score >2), aneurysms, ectasia, pericardial effusion requiring drainage, or focal wall abnormalities suggestive of myocardial ischemia
13. Chest tube
14. Concurrent dialysis
15. Suspected CNS infection
16. Severe bronchospasm requiring continuous bronchodilators
17. Pulmonary hemorrhage
18. A formal diagnosis of full Kawasaki disease (KD).
19. Failure to perform COVID-19 PCR and serology testing prior to IVIG administration.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the Investigational Product, hCT-MSCs, infusion reactions | 2 days post infusion
  Incidence of infusion reactions
Safety of the Investigational Product, hCT-MSCs, related adverse events | 90 days post initial infusion
  Incidence of later reactions attributed to the investigational product
Safety of the Investigational Product, hCT-MSCs, anti-HLA antibodies | from first dose of MSCs to 28 days after first dose
  Incidence of formation of new anti-HLA antibodies post infusion as compared to pre-infusion levels.

SECONDARY OUTCOMES:
Survival | from first dose of MSCs to 28 days after first dose
  Survival rate at 28 days after the first dose of MSCs
Inotrope support | from first dose of MSCs to 90 days after first dose
  Description of duration of inotrope support after the first dose of MSCs
Hospital Discharge | from first dose of MSCs to 90 days after first dose
  Description of number of days to hospital discharge to home
Duration of ICU stay | from first dose of MSCs to 90 days after first dose
  Description of Duration of ICU stay
cardiac abnormalities | from first dose of MSCs to 28 days after first dose
  Incidence of cardiac abnormalities at day 28, defined as persistent abnormalities in ECG, Echo, or biochemical markers (pro-BNP, troponin).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - New York Medical College, Westchester Medical Center (WMC), Westchester, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No